CLINICAL TRIAL: NCT04843761
Title: A Multicenter, Adaptive, Randomized, Blinded Controlled Trial of the Safety and Efficacy of Investigational Therapeutics for Hospitalized Patients With Acute Respiratory Distress Syndrome Associated With COVID-19
Brief Title: ACTIV-3b: Therapeutics for Severely Ill Inpatients With COVID-19
Acronym: TESICO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: International Network for Strategic Initiatives in Global HIV Trials (INSIGHT) (Network); University of Copenhagen (Other); Medical Research Council (Other Government); Kirby Institute (Other Government); Washington D.C. Veterans Affairs Medical Center (U.S. Federal Agency); Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections (Network); US Department of Veterans Affairs (U.S. Federal Agency); Prevention and Early Treatment of Acute Lung Injury (PETAL) Network (Unknown); NeuroRx, Inc. (Industry); Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 015 / ACTIV-3b
Record Dates: First submitted 2021-04-09; First posted 2021-04-14 (Actual); Results first posted 2025-10-24 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-09

CONDITIONS: Covid19
Keywords: COVID-19; COVID 19; Coronaviridae Infections; Coronavirus Infections; RNA Virus Infections; Virus Diseases; Nidovirales Infections; SARS-CoV-2; SARS Coronavirus; ACTIV-3; ACTIV3
MeSH Terms: conditions — COVID-19; Coronaviridae Infections; Coronavirus Infections; RNA Virus Infections; Virus Diseases; Nidovirales Infections; Severe Acute Respiratory Syndrome | interventions — remdesivir; aviptadil; Vasoactive Intestinal Peptide; Adrenal Cortex Hormones

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- Stratum 1 - Aviptadil + Remdesivir + SOC (Experimental): Eligible for both Aviptadil and Remdesivir and no prior use of Remdesivir
  Participants enrolled in Stratum 1 were analyzed in both substudies (H1: NCT06729606; H2: NCT06729593)
  Interventions: Biological: Remdesivir; Biological: Aviptadil; Drug: Corticosteroid
- Stratum 1 - Aviptadil + Remdesivir Placebo + SOC (Experimental): Eligible for both Aviptadil and Remdesivir and no prior use of Remdesivir
  Participants enrolled in Stratum 1 were analyzed in both substudies (H1: NCT06729606; H2: NCT06729593)
  Interventions: Drug: Remdesivir Placebo; Biological: Aviptadil; Drug: Corticosteroid
- Stratum 1 - Aviptadil Placebo + Remdesivir + SOC (Experimental): Eligible for both Aviptadil and Remdesivir and no prior use of Remdesivir
  Participants enrolled in Stratum 1 were analyzed in both substudies (H1: NCT06729606; H2: NCT06729593)
  Interventions: Biological: Remdesivir; Drug: Aviptadil Placebo; Drug: Corticosteroid
- Stratum 1 - Aviptadil Placebo + Remdesivir Placebo + SOC (Placebo Comparator): Eligible for both Aviptadil and Remdesivir and no prior use of Remdesivir
  Participants enrolled in Stratum 1 were analyzed in both substudies (H1: NCT06729606; H2: NCT06729593)
  Interventions: Drug: Remdesivir Placebo; Drug: Aviptadil Placebo; Drug: Corticosteroid
- Stratum 2 - Aviptadil + SOC (Experimental): Eligible for Aviptadil and Remdesivir contraindicated
  * Contraindications: eGFR less than 30 or ALT/AST greater than 10x the upper limit of normal
  Participants enrolled in this arm were analyzed in substudy H1 (NCT06729606)
  Interventions: Biological: Aviptadil; Drug: Corticosteroid
- Stratum 2 - Aviptadil Placebo + SOC (Placebo Comparator): Eligible for Aviptadil and Remdesivir contraindicated
  * Contraindications: eGFR less than 30 or ALT/AST greater than 10x the upper limit of normal
  Participants enrolled in this arm were analyzed in substudy H1 (NCT06729606)
  Interventions: Drug: Aviptadil Placebo; Drug: Corticosteroid
- Stratum 3 - Remdesivir + SOC (Experimental): Eligible for Remdesivir and Aviptadil contraindicated
  * Contraindications: refractory hypotension (norepinephrine equivalent greater than or equal to 0.1 mcg/kg/min), severe diarrhea, end-stage liver disease, c-diff infection
  Participants enrolled in this arm were analyzed in substudy H2 (NCT06729593)
  Interventions: Biological: Remdesivir; Drug: Corticosteroid
- Stratum 3 - Remdesivir Placebo + SOC (Placebo Comparator): Eligible for Remdesivir and Aviptadil contraindicated
  * Contraindications: refractory hypotension (norepinephrine equivalent greater than or equal to 0.1 mcg/kg/min), severe diarrhea, end-stage liver disease, c-diff infection
  Participants enrolled in this arm were analyzed in substudy H2 (NCT06729593)
  Interventions: Drug: Remdesivir Placebo; Drug: Corticosteroid
- Stratum 4 - Aviptadil + SOC (Experimental): Eligible for Aviptadil and prior/current use of Remdesivir
  Participants enrolled in this arm were analyzed in substudy H1 (NCT06729606)
  Interventions: Biological: Aviptadil; Drug: Corticosteroid
- Stratum 4 - Aviptadil Placebo + SOC (Placebo Comparator): Eligible for Aviptadil and prior/current use of Remdesivir
  Participants enrolled in this arm were analyzed in substudy H1 (NCT06729606)
  Interventions: Drug: Aviptadil Placebo; Drug: Corticosteroid

INTERVENTIONS:
Biological: Remdesivir — Administered by IV infusion, daily for 10 days. Initial loading dose is 200 mg with all subsequent doses 100 mg.
  Arms: Stratum 1 - Aviptadil + Remdesivir + SOC; Stratum 1 - Aviptadil Placebo + Remdesivir + SOC; Stratum 3 - Remdesivir + SOC
Drug: Remdesivir Placebo — Commercially available 0.9% sodium chloride solution. Administered by IV infusion daily for 10 days.
  Arms: Stratum 1 - Aviptadil + Remdesivir Placebo + SOC; Stratum 1 - Aviptadil Placebo + Remdesivir Placebo + SOC; Stratum 3 - Remdesivir Placebo + SOC
Biological: Aviptadil — Administered by IV infusion over 12 hours per day for 3 days. The Day 1 infusion rate is 50 pmol/kg/hr, the Day 2 infusion rate is 100 pmol/kg/hr, and the Day 3 infusion rate is 150 pmol/kg/hr.
  Other Names: Vasoactive Intestinal Peptide; VIP
  Arms: Stratum 1 - Aviptadil + Remdesivir + SOC; Stratum 1 - Aviptadil + Remdesivir Placebo + SOC; Stratum 2 - Aviptadil + SOC; Stratum 4 - Aviptadil + SOC
Drug: Aviptadil Placebo — Commercially available 0.9% sodium chloride solution. Administered by IV infusion over 12 hours per day for 3 days.
  Arms: Stratum 1 - Aviptadil Placebo + Remdesivir + SOC; Stratum 1 - Aviptadil Placebo + Remdesivir Placebo + SOC; Stratum 2 - Aviptadil Placebo + SOC; Stratum 4 - Aviptadil Placebo + SOC
Drug: Corticosteroid — In line with NIH treatment guidelines, corticosteroids such as dexamethasone, prednisone, methylprednisolone or hydrocortisone may be administered as SOC.

SUMMARY:
This study looks at the safety and effectiveness of different drugs in treating COVID-19 in people who have been hospitalized with the infection and who have acute respiratory failure. Participants in the study will be treated with either a study drug plus current standard of care (SOC), or with placebo plus current SOC.

Substudy H1: Aviptadil for Severely Ill Inpatients With COVID-19 (NCT06729606)

Substudy H2: Remdesivir for Severely Ill Inpatients With COVID-19 (NCT06729593)

DETAILED DESCRIPTION:
This is a master protocol to evaluate the safety and efficacy of investigational agents aimed at improving outcomes for patients with acute respiratory failure related to COVID-19.

Trials within this protocol will be adaptive, randomized, blinded and initially placebo-controlled. Participants will receive standard of care (SOC) treatment as part of the protocol. If an investigational agent shows superiority over placebo, SOC for the study of future investigational agents may be modified accordingly.

The international trials within this protocol will be conducted in up to several hundred clinical sites. Participating sites are affiliated with networks funded by the United States National Institutes of Health (NIH) and the US Department of Veterans Affairs.

The protocol is for a Phase 3 platform study that allows investigational agents to be added and dropped during the course of the study. This allows for efficient testing of new agents against control within the same trial infrastructure. When more than one agent is being tested concurrently, participants may be randomly allocated across agents (as well as between the agent and its placebo) so the same control group can be shared, when feasible. In some situations, a factorial design may be used to study multiple agents.

Participants will be followed for 90 days following randomization for the primary endpoint and most secondary endpoints. Selected secondary endpoints will be measured at 180 days.

This study is planned to provide 80% power to detect an odds ratio of 1.5 for improvement in recovery status at Day 90 for an investigational agent versus placebo with use of the ordinal outcome. The planned sample size is 640 participants (320 per group) for each investigational agent/placebo. Sample size may be re-estimated before enrollment is complete based on an assessment of whether the pooled proportions of the outcome are still consistent with adequate power for the hypothesized difference measured by the odds ratio.

Randomization will be stratified by study site pharmacy and by receipt of invasive mechanical ventilation, or ECMO (extracorporeal membrane oxygenation) at enrollment. Other agent-specific stratification factors may be considered.

Investigational agents suitable for testing in the inpatient setting will be prioritized based on in vitro data, preclinical data, Phase 1 pharmacokinetic and safety data, and clinical data from completed and ongoing trials. In some cases, a vanguard cohort/initial pilot phase may be incorporated into the trial.

An independent Data and Safety Monitoring Board (DSMB) will review interim safety and efficacy data at least monthly. Pre-specified guidelines will be established to recommend early stopping of the trial for evidence of harm or substantial efficacy. The DSMB may recommend discontinuation of an investigational agent if the risks are judged to outweigh the benefits.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent.
* Requiring admission for inpatient hospital acute medical care for clinical manifestations of COVID-19 (not for purely public health or quarantine purposes).
* Current respiratory failure (i.e. receipt of high-flow nasal cannula, non-invasive ventilation, invasive mechanical ventilation, or ECMO used to treat acute hypoxemic respiratory failure).
* SARS-CoV-2 (COVID-19) infection, documented by a nucleic acid test (NAT) or equivalent testing with most recent rest within 14 days prior to randomization.
* Respiratory failure is believed to be due to SARS-CoV-2 pneumonia.

Exclusion Criteria:

* Known allergy to investigational agent or vehicle.
* More than 4 days since initiation of support for respiratory failure.
* Chronic/home mechanical ventilation (invasive or non-invasive) for chronic lung or neuromuscular disease (non-invasive ventilation used solely for sleep-disordered breathing is not an exclusion).
* Moribund patient (i.e. not expected to survive 24 hours).
* Active use of "comfort care" or other hospice-equivalent SOC.
* Expected inability to participate in study procedures.
* In the opinion of the investigator, any condition for which, participation would not be in the best interest of the participant or that could limit protocol-specified assessments.
* Previous enrollment in TESICO

Additional agent-specific criteria also apply, and are listed in the substudy records Substudy H1: Aviptadil for Severely Ill Inpatients With COVID-19 (NCT06729606) Substudy H2: Remdesivir for Severely Ill Inpatients With COVID-19 (NCT06729593)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 473 (Actual)
Dates: Start 2021-04-20 (Actual); Primary Completion 2022-08-22 (Actual); Study Completion 2022-11-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Brown, MD, Principal Investigator — Intermountain Medical Center/University of Utah; Prof. James Neaton, Study Chair — INSIGHT Statistical and Coordinating Centre, University of Minnesota
Locations (40):
- United States (40):
  - Banner University Medical Center Tucson (Site 206-004), 1625 N. Campbell Avenue, Tucson, Arizona
  - UCSF Fresno (Site 203-005), 155 N. Fresno Street, Fresno, California
  - VA Loma Linda Healthcare System (Site 074-017), 11201 Benton Street, Loma Linda, California
  - Cedars-Sinai Medical Center (Site 208-002), 8700 Beverly Boulevard, Los Angeles, California
  - Ronald Reagan UCLA Medical Center (Site 203-002), 757 Westwood Plaza, Los Angeles, California
  - UCSF Medical Center at Mount Zion (Site 203-007), 1600 Divisadero St., San Francisco, California
  - UCSF Medical Center (Site 203-001), Moffit-Long Hospital, 505 Parnassus Ave., San Francisco, California
  - Stanford University Hospital & Clinics (Site 203-003), 300 Pasteur Dr., Stanford, California
  - University of Colorado Hospital (Site 204-001), 12605 E. 16th Avenue, Aurora, Colorado
  - Denver Health Medical Center (Site 204-004), 780 Delaware Street, Pavilion B, Denver, Colorado
  - MedStar Health Research Institute (Site 009-021), 110 Irving St., NW., Washington D.C., District of Columbia
  - Washington DC VA Medical Center (Site 009-004), 50 Irving Street, NW., Washington D.C., District of Columbia
  - Emory University (Site 301-008), Bldg. A, Suite 2236, 1365 Clifton Rd., NE., Atlanta, Georgia
  - Massachusetts General Hospital (Site 202-002), 55 Fruit Street, Boston, Massachusetts
  - Baystate Medical Center (Site 201-001), Critical Care Research, 759 Chestnut Street, Springfield, Massachusetts
  - Mount Sinai Medical Center (Site 301-012), Icahn School of Medicine at Mount Sinai, One Gustave L. Levy Place, New York, New York
  - Columbia University Irving Medical Center (Site 301-027), 177 Fort Washington Ave., New York, New York
  - Montefiore Medical Center - Moses Hospital (Site 206-001), 111 E. 210th Street, The Bronx, New York
  - Montefiore Medical Center - Weiler campus (Site 206-003), 111 E. 210th Street, The Bronx, New York
  - Duke University Hospital (Site 301-006), 2301 Erwin Road, Durham, North Carolina
  - Wake Forest Baptist Health (Site 210-001), Medical Center Blvd, Winston-Salem, North Carolina
  - University of Cincinnati Medical Center (Site 207-003), 234 Goodman Street, ML 0740, Cincinnati, Ohio
  - Cleveland Clinic Fairview Hospital (Site 207-005), 18101 Lorain Ave., Cleveland, Ohio
  - Cleveland Clinic Foundation (Site 207-001), 9500 Euclid Ave., Cleveland, Ohio
  - The Ohio State University Wexner Medical Center (Site 207-004), 410 W. 10th Avenue, Columbus, Ohio
  - Cleveland Clinic Marymount Campus (Site 207-006), 12300 McCracken Road, Garfield Heights, Ohio
  - Cleveland Clinic Hillcrest Hospital (Site 207-007), 6780 Mayfield Road, Mayfield Heights, Ohio
  - Oregon Health & Science University (Site 208-003), 3181 SW Sam Jackson Park Rd., Portland, Oregon
  - Medical University of South Carolina (Site 210-002), 96 Jonathan Lucas St., CSB 214, Charleston, South Carolina
  - Vanderbilt University Medical Center (Site 212-001), 1211 Medical Center Drive, Nashville, Tennessee
  - Baylor, Scott and White Health (Site 301-003), Baylor University Medical Center, 3500 Gaston Ave., Dallas, Texas
  - Houston Methodist Hospital (Site 301-028), 6565 Fannin Street, Houston, Texas
  - Texas Heart Institute (Site 301-017), 6770 Bertner, MC4-266, Houston, Texas
  - University of Texas Health Science Center (Site 203-006), 7000 Fannin St., Houston, Texas
  - Intermountain Medical Center (Site 211-001), 5121 South Cottonwood Street, Murray, Utah
  - University of Utah Hospital (Site 211-002), 50 North Medical Drive, Salt Lake City, Utah
  - UVA School of Medicine (Site 210-003), University of Virginia Health System, University Hospital, 1215 Lee St., Charlottesville, Virginia
  - Harborview Medical Center (Site 208-001), 325 9th Ave., Seattle, Washington
  - Swedish Medical Center (Site 208-005), 747 Broadway, Seattle, Washington
  - West Virginia University Medicine (Site 301-023), One Medical Center Drive, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Brown SM, Barkauskas CE, Grund B, Sharma S, Phillips AN, Leither L, Peltan ID, Lanspa M, Gilstrap DL, Mourad A, Lane K, Beitler JR, Serra AL, Garcia I, Almasri E, Fayed M, Hubel K, Harris ES, Middleton EA, Barrios MAG, Mathews KS, Goel NN, Acquah S, Mosier J, Hypes C, Salvagio Campbell E, Khan A, Hough CL, Wilson JG, Levitt JE, Duggal A, Dugar S, Goodwin AJ, Terry C, Chen P, Torbati S, Iyer N, Sandkovsky US, Johnson NJ, Robinson BRH, Matthay MA, Aggarwal NR, Douglas IS, Casey JD, Hache-Marliere M, Georges Youssef J, Nkemdirim W, Leshnower B, Awan O, Pannu S, O'Mahony DS, Manian P, Awori Hayanga JW, Wortmann GW, Tomazini BM, Miller RF, Jensen JU, Murray DD, Bickell NA, Zatakia J, Burris S, Higgs ES, Natarajan V, Dewar RL, Schechner A, Kang N, Arenas-Pinto A, Hudson F, Ginde AA, Self WH, Rogers AJ, Oldmixon CF, Morin H, Sanchez A, Weintrob AC, Cavalcanti AB, Davis-Karim A, Engen N, Denning E, Taylor Thompson B, Gelijns AC, Kan V, Davey VJ, Lundgren JD, Babiker AG, Neaton JD, Lane HC; ACTIV-3b/Therapeutics for Severely Ill Inpatients with COVID-19 (TESICO) Study Group. Intravenous aviptadil and remdesivir for treatment of COVID-19-associated hypoxaemic respiratory failure in the USA (TESICO): a randomised, placebo-controlled trial. Lancet Respir Med. 2023 Sep;11(9):791-803. doi: 10.1016/S2213-2600(23)00147-9. Epub 2023 Jun 19. PMID 37348524
- [Derived] Grundeis F, Ansems K, Dahms K, Thieme V, Metzendorf MI, Skoetz N, Benstoem C, Mikolajewska A, Griesel M, Fichtner F, Stegemann M. Remdesivir for the treatment of COVID-19. Cochrane Database Syst Rev. 2023 Jan 25;1(1):CD014962. doi: 10.1002/14651858.CD014962.pub2. PMID 36695483
- [Derived] Tsiatis AA, Davidian M, Holloway ST. Estimation of the odds ratio in a proportional odds model with censored time-lagged outcome in a randomized clinical trial. Biometrics. 2023 Jun;79(2):975-987. doi: 10.1111/biom.13603. Epub 2021 Dec 17. PMID 34825704
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm
- See also: CDC (Centers for Disease Control and Prevention): Coronavirus (COVID-19) website — https://www.cdc.gov/coronavirus/2019-nCoV/index.html
- See also: A Participant's Guide to Clinical Trials (NIAID) — https://www.niaid.nih.gov/clinical-trials/participant-guide
- See also: Find a Clinical Trial (NIAID) — https://www.niaid.nih.gov/clinical-trials/find-a-clinical-trial
- See also: Clinical Trials at NIAID — https://www.niaid.nih.gov/clinical-trials
- See also: National Institute for Allergy and Infectious Diseases (NIAID) — https://www.niaid.nih.gov/
- See also: WHO COVID-19 treatment guidelines — https://www.who.int/emergencies/diseases/novel-coronavirus-2019/technical-guidance/patient-management

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligibility for each agent was assessed at the same time.
  If eligible for both, participants were randomized to a 2x2 factorial design of Aviptadil vs. Aviptadil placebo and Remdesivir vs. Remdesivir placebo with 1:1:1:1 allocation to each of the 4 possible combinations. If eligible for only 1, randomization was 1:1 to that agent or its matched placebo (Appendix H2).
  The primary analysis for each agent was to pool across applicable groups to compare each agent vs. matched placebo.
Pre-assignment Details: The study includes randomization according to 4 strata:
  * Stratum 1 eligible for both Aviptadil and Remdesivir (no prior Remdesivir)
  * Stratum 2 eligible for Aviptadil only (Remdesivir contraindicated)
  * Stratum 3 eligible for Remdesivir only (Aviptadil contraindicated)
  * Stratum 4 eligible for Aviptadil and have received prior Remdesivir
  This record presents enrollment data across the full study. Refer to the agent-specific records for results by agent (H1: NCT06729606; H2: NCT06729593)
Groups:
- Stratum 1 - Aviptadil + Remdesivir; Stratum 1 - Aviptadil +Remdesivir Placebo; Stratum 1 - Aviptadil Placebo + Remdesivir; Stratum 1 - Aviptadil Placebo + Remdesivir Placebo: Eligible for both Aviptadil and Remdesivir and no prior use of Remdesivir
  * Participants enrolled in Stratum 1 were analyzed in both substudies (H1: NCT06729606; H2: NCT06729593)
- Stratum 2 - Aviptadil; Stratum 2 - Aviptadil Placebo: Eligible for Aviptadil and Remdesivir contraindicated
  * Contraindications: eGFR less than 30 or ALT/AST greater than 10x the upper limit of normal
  * Participants enrolled in this arm were analyzed in substudy H1 (NCT06729606)
- Stratum 3 - Remdesivir; Stratum 3 - Remdesivir Placebo: Eligible for Remdesivir and Aviptadil contraindicated
  * Contraindications: refractory hypotension (norepinephrine equivalent greater than or equal to 0.1 mcg/kg/min), severe diarrhea, end-stage liver disease, c-diff infection
  * Participants enrolled in this arm were analyzed in substudy H2 (NCT06729593)
- Stratum 4 - Aviptadil; Stratum 4 - Aviptadil Placebo: Eligible for Aviptadil and prior/current use of Remdesivir
  * Participants enrolled in this arm were analyzed in substudy H1 (NCT06729606)
Period: Overall Study
Arm/Group | Stratum 1 - Aviptadil + Remdesivir | Stratum 1 - Aviptadil +Remdesivir Placebo | Stratum 1 - Aviptadil Placebo + Remdesivir | Stratum 1 - Aviptadil Placebo + Remdesivir Placebo | Stratum 2 - Aviptadil | Stratum 2 - Aviptadil Placebo | Stratum 3 - Remdesivir | Stratum 3 - Remdesivir Placebo | Stratum 4 - Aviptadil | Stratum 4 - Aviptadil Placebo
Started | 18 | 21 | 25 | 21 | 12 | 11 | 1 | 1 | 183 | 180
Completed | 18 | 21 | 25 | 21 | 12 | 11 | 1 | 1 | 183 | 180
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Stratum 1 - Aviptadil + Remdesivir | Stratum 1 - Aviptadil +Remdesivir Placebo | Stratum 1 - Aviptadil Placebo + Remdesivir | Stratum 1 - Aviptadil Placebo + Remdesivir Placebo | Stratum 2 - Aviptadil | Stratum 2 - Aviptadil Placebo | Stratum 3 - Remdesivir | Stratum 3 - Remdesivir Placebo | Stratum 4 - Aviptadil | Stratum 4 - Aviptadil Placebo | Total
Number analyzed (Participants) | 18 | 21 | 25 | 21 | 12 | 11 | 1 | 1 | 183 | 180 | 473
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (13) | 55 (14) | 56 (15) | 56 (11) | 60 (20) | 54 (21) | 71 (0) | 70 (0) | 57 (15) | 57 (15) | 57 (15)
Age, Customized [Count of Participants; unit: Participants]
  <= 18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 15 | 14 | 14 | 17 | 6 | 7 | 0 | 0 | 123 | 126 | 322
  >= 65 years | 3 | 7 | 11 | 4 | 6 | 4 | 1 | 1 | 60 | 54 | 151
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 8 | 7 | 9 | 2 | 1 | 1 | 74 | 71 | 185
  Male | 13 | 14 | 17 | 14 | 3 | 9 | 0 | 0 | 109 | 109 | 288
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 7 | 7 | 9 | 3 | 3 | 1 | 0 | 46 | 40 | 122
  Not Hispanic or Latino | 12 | 14 | 18 | 12 | 9 | 8 | 0 | 1 | 137 | 140 | 351
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 7
  Asian | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 5 | 9 | 17
  Native Hawaiian or Pacific Islander | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 3 | 1 | 6
  Black or African American | 3 | 2 | 3 | 2 | 2 | 1 | 0 | 0 | 33 | 27 | 73
  White | 6 | 13 | 12 | 10 | 6 | 9 | 1 | 1 | 101 | 107 | 266
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Other | 1 | 2 | 2 | 0 | 2 | 1 | 0 | 0 | 11 | 9 | 28
  Only ethnicity (race unknown) | 6 | 3 | 6 | 7 | 2 | 0 | 0 | 0 | 29 | 23 | 76

OUTCOME MEASURES:

1. Primary Outcome: Substudy Analysis Cohorts
Description: The primary analysis for each agent was to pool across applicable groups to compare each agent vs. matched placebo. Refer to the agent-specific records for results by agent (H1 [Aviptadil]: NCT06729606; H2 [Remdesivir]: NCT06729593).
Time Frame: Screening, within 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Stratum 1 - Aviptadil + Remdesivir | Stratum 1 - Aviptadil +Remdesivir Placebo | Stratum 1 - Aviptadil Placebo + Remdesivir | Stratum 1 - Aviptadil Placebo + Remdesivir Placebo | Stratum 2 - Aviptadil | Stratum 2 - Aviptadil Placebo | Stratum 3 - Remdesivir | Stratum 3 - Remdesivir Placebo | Stratum 4 - Aviptadil | Stratum 4 - Aviptadil Placebo
Number analyzed (Participants) | 18 | 21 | 25 | 21 | 12 | 11 | 1 | 1 | 183 | 180
Participants
  Aviptadil substudy analysis cohort | 18 | 21 | 25 | 21 | 12 | 11 | 0 | 0 | 183 | 180
  Remdesivir substudy analysis cohort | 18 | 21 | 25 | 21 | 0 | 0 | 1 | 1 | 0 | 0

ADVERSE EVENTS:
Time Frame: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed during the screening phase of the study
Description: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed during the screening phase of the study
Arm/Group | Stratum 1 - Aviptadil + Remdesivir | Stratum 1 - Aviptadil +Remdesivir Placebo | Stratum 1 - Aviptadil Placebo + Remdesivir | Stratum 1 - Aviptadil Placebo + Remdesivir Placebo | Stratum 2 - Aviptadil | Stratum 2 - Aviptadil Placebo | Stratum 3 - Remdesivir | Stratum 3 - Remdesivir Placebo | Stratum 4 - Aviptadil | Stratum 4 - Aviptadil Placebo
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (7):
  • Study Protocol: Master (2022-03-08): https://cdn.clinicaltrials.gov/large-docs/61/NCT04843761/Prot_008.pdf
  • Study Protocol: Aviptadil (H1) (2022-03-08): https://cdn.clinicaltrials.gov/large-docs/61/NCT04843761/Prot_009.pdf
  • Study Protocol: Remdesivir (H2) (2021-04-01): https://cdn.clinicaltrials.gov/large-docs/61/NCT04843761/Prot_010.pdf
  • Study Protocol: Overview of Study Documents (2025-08-05): https://cdn.clinicaltrials.gov/large-docs/61/NCT04843761/Prot_011.pdf
  • Statistical Analysis Plan: Main (2021-08-05): https://cdn.clinicaltrials.gov/large-docs/61/NCT04843761/SAP_012.pdf
  • Statistical Analysis Plan: Addendum (2022-05-01): https://cdn.clinicaltrials.gov/large-docs/61/NCT04843761/SAP_013.pdf
  • Informed Consent Form (2022-03-08): https://cdn.clinicaltrials.gov/large-docs/61/NCT04843761/ICF_014.pdf